CLINICAL TRIAL: NCT05089955
Title: User Evaluation New Ambient Experience Content
Brief Title: Children's MRI Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ICBE-S-000195
Record Dates: First submitted 2021-09-10; First posted 2021-10-22 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Behavior; Psychological Distress; Anxiety
MeSH Terms: conditions — Behavior; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): MRI examination with Ambient Experience with paediatric content
  Interventions: Behavioral: Ambient Experience
- Control group (No Intervention): MRI examination without Ambient Experience (standard of care)

INTERVENTIONS:
Behavioral: Ambient Experience — MRI examination with Ambient Experience
  Arms: Intervention group

SUMMARY:
The study aims to investigate the effect of Philips Ambient Experience with specially designed paediatric content on the experience of pediatric patients undergoing an MRI examination, their caregiver, and clinical staff, on workflow and on clinical outcome. The designed paediatric content exists of personal selection of a character, video projection on the wall and/or a screen visible when in the bore, audio, and room ambience lighting.

The study will be conducted in collaboration with six partner hospitals within the EU. At each hospital, 50 pediatric patients between 6 and 12 years old will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 6 and 12 years old
* Scheduled for a head-first MRI scan
* Parent/guardian and child speak and read the local language.
* Positive judgement by on-site PI/(co-) investigator for awake scanning

Exclusion Criteria:

* General anesthesia
* Clinically diagnosed cognitive, or developmental disorder (e.g. ADHD, ASD) or neurological problems that prevent the ability to lie/hold still for an MRI scan while awake
* Previous MRI examination with Philips Ambient Experience

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Child anxiety level | The visit on the imaging department; before and after the examination. This is estimated to be 30 up to 60 minutes, depending on the MRI scans that have to be made.
  Change of anxiety experienced by the child, measured with questions before and after the scan. A Venham picture preference scale will be used, the range is not applicable as it indicates their state of anxiety.
Child anxiety level | The visit on the imaging department; before and during the examination. This is estimated to be 10 up to 30 minutes, depending on the MRI scans that have to be made.
  Change of anxiety level of child measured with an observational scale by staff or (co-) investigator before and during the scan. By using a modified yale preoperative anxiety scale, with a range from 22.92 to 100; higher values indicating greater anxiety.

SECONDARY OUTCOMES:
Immersiveness and engagement with Ambient Experience and content | After the scan, 5 minutes.
  Measured with likability of the experience and characters. This scale is self-constructed for the purpose of measuring how much the child likes the characters and how much that influenced their experience of the scan.
Parent/ Guardian satisfaction | After the scan, 5 minutes
  Will be measured with self-constructed 6-point Likert scale, with higher ratings indicating a higher satisfaction.

OTHER OUTCOMES:
Staff experience with the ambient experience system and workflow satisfaction | At study start 5 min. and study end 5 min.
  Measured by using self-constructered items, 5 point Likert scales, with higher ratings indicating a better experience and higher satisfaction.
Observed operational efficiency | 5 minutes depending on the MRI scans that have to be made
  Observed cooperation of the patient and duration of preparing the patient for the MRI examination.This will be measured by using 5-point Likert scales, with higher ratings indicating a lower efficiency.
Measured operational efficiency | 30 up to 60 minutes depending on the entire length of the MRI scans that have to be made
  Duration of the MRI examination, number of rescans required, and number of pauzes required. Numerical log data derived from the MRI server.
Clinical patient outcome | During MRI scan, ca 30 minutes
  Reported image quality by the MRI tech and the ability to perform the planned awake scan successful or not

CONTACTS AND LOCATIONS:
Overall Officials: Sanae van der Vleuten- Chraibi, Study Director — Philips Electronics Nederland B.V. acting through Philips CTO organization
Locations (6):
- UZ Brussel, Jette, Brussels Capital, Belgium
- Herlev Hospital, Herlev, Denmark
- Hôpital Robert Debré Paris, Paris, France
- Das Universitätsklinikum Bonn (UKB), Bonn, North Rhine-Westphalia, Germany
- Polish Mother's Hospital / Institute of Polish Mother's Health Center, Lodz, Poland
- Hospital de Sant Joan de Déu Barcelona, Esplugues de Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] van der Vleuten-Chraibi S, Nauts S, Baranska D, Inarejos Clemente EJ, Sterup Bovin J, Najafi N, Luetkens JA, Alison M, Biermann HM, Peckman F, Saini P. Magnetic resonance imaging related anxiety and workflow: impact of a child-friendly audio-visual intervention. Pediatr Radiol. 2025 Aug;55(9):1934-1942. doi: 10.1007/s00247-025-06308-0. Epub 2025 Jul 4. PMID 40613840